CLINICAL TRIAL: NCT00469664
Title: A Double Blind Placebo Controlled Study of Guanfacine Adjunctive Treatment to Atypical Antipsychotics for Cognitive Dysfunction in Schizophrenia
Brief Title: Guanfacine Adjunctive Treatment to Atypical Antipsychotics for Cognitive Dysfunction in Schizophrenia
Acronym: Guanfacine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Bronx VA Medical Center (U.S. Federal Agency); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Joseph Friedman, MD, PilgrimPsychiatric Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00110; 99-621
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Cognitive Impairment
Keywords: Schizophrenia; Schizoaffective; Cognitive Impairment; Cognition; Memory; Attention; Concentration
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognitive Dysfunction | interventions — Guanfacine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Guanfacine/Tenex

SUMMARY:
Our overall aim is to determine if the administration of guanfacine in combination with aripiprazole, olanzapine, quetiapine, and/or risperidone is significantly more effective than any of those medications alone in treating some of the cognitive impairment in schizophrenia.

DETAILED DESCRIPTION:
The proposed study is a double blind, placebo controlled, parallel designed investigation comparing the effect of one of four atypical antipsychotics (aripiprazole, olanzapine, quetiapine, and/or risperidone), treatment alone to treatment with one of these in addition to treatment with guanfacine to maximum dose of 3.0 mg per day on a cognitive task performance in schizophrenic patients. The study will take place over fourteen weeks. Patients will receive study medication for the last ten weeks of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males and females between the ages of 18 and 55.
2. In good general medical health.
3. Have a DSMIV diagnosis of schizophrenia, any subtype, or schizoaffective disorder.
4. Patients who have been diagnosed with other DSMIV Axis I disorders may be included, unless they are actively using illicit substances.
5. Receiving treatment with aripiprazole, olanzapine, quetiapine, and/or risperidone as their antipsychotic medication
6. Subjects will demonstrate significant memory impairment by performing at least two standard deviations below normal performance on the California Verbal Learning Test (CVLT). Using subjects with a clear impairment in acquisition and recall will avoid a ceiling effect in this measure.
7. Subjects will also be required to have at least an 8th grade reading level and/or a full-scale IQ of at least 85 as assessed by the Wide Range Achievement Test (WRAT).
8. Patients are allowed to be on the following anti-depressant medications: Fluoxetine (PROZAC), Sertraline (ZOLOFT), Paroxetine (PAXIL), Celexa (CITALOPRAM), Busprion (WELLBUTRIN), Venlafaxine (EFFEXOR), and Buspirone (BUSPAR).

Exclusion Criteria:

1. Have a recent history (within previous year) of serious suicide, homicide, or serious physical violence, or current suicidal or homicidal thoughts
2. Active use of illicit substances.
3. Meet DSM-IV criteria for a current episode of major depression or mania.
4. Have a history of severe head trauma, neurological disorder or medical illness which may contribute to the patient's psychiatric symptoms and cognitive impairment.
5. Have a medical illness which requires that they take any medication that has CNS activity or which is known to interact with guanfacine (e.g barbiturates, apha-1 antagonists, beta blockers).
6. Receive treatment with other concomitant neuroleptics in addition to risperidone or olanzapine.
7. Receive concomitant anticholinergic drugs, or. If the patient receives benzodiazepines, they must be short or intermediate acting (e.g. alprazolam, lorazepam) and they must be held 48 hours prior to cognitive testing. Treatment with mood stabilizers such as lithium and depakote will be allowed for this study. If the patients is receiving treatment with lithium the level must be < 1 meq/l.
8. Are unable to give informed consent.
9. Have a history of developmental disorder or less than an eighth grade reading level.
10. Have a history of bowel obstruction or untreated benign prostatic hypertrophy. Are taking antihypertensive medications of the class of beta-blockers, alpha-1 antagonists, calcium channel blockers, or alpha-2 agonists.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2000-02; Primary Completion 2008-08 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Spatial Working Memory Test Trail Making Test: Part A and B. | Baseline, week 6, week 10

SECONDARY OUTCOMES:
RAVLT,Digit Span Distraction Test,CPT450,Verbal Fluency Test, Wisconsin Card Sorting Test,Stroop Interference Test,Letter-Number Sequencing, Extra Pyramidal Symptom Rating Scale(ESRS),Positive And Negative Symptom Scale | Baseline, week 6, week 10

CONTACTS AND LOCATIONS:
Overall Officials: Joseph I Friedman, MD, Principal Investigator — Pilgrim Psychiatric Center, Mount Sinai Medical Center, Bronx VA Medical Center
Locations (3):
- United States (3):
  - Mount Sinai Medical Center, New York, New York
  - Bronx VA Medical Center, The Bronx, New York
  - Pilgrim Psychiatric Center, W. Brentwood, New York